CLINICAL TRIAL: NCT05669378
Title: A Good Start Matters: Do Supportive Childcare Centre Environments, Policies and Practices Enhance Physical Activity?
Brief Title: A Good Start Matters Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Louise Masse, Professor and Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H18-01434
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Physical Inactivity; Motor Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: To test the efficacy of ATP+, we will conduct a randomized control trial with 52 facilities - where 26 facilities will be randomized to receive the intervention and while the remaining facilities will receive the standard of care as a waitlist control group and will receive the intervention at 3-month post randomization.
Who Masked: Outcomes Assessor
Masking Description: Partial masking as the outcome assessors will not deliver intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will receive the Appetite to Play + intervention which is a capacity-building intervention that support childcare providers in implementing the best practices for active play. It includes a 3 e-learning online modules and then the are supported with weekly . bi-weekly emails.
  Interventions: Behavioral: Appetite to Play +
- Standard of care waitlist control (Other): The standard of care waitlist control group will receive the intervention at 3-months post-randomization. The standard of care group has access to the Appetite to Play materials which are available to everyone. The site includes resources that childcare providers can use.
  Interventions: Behavioral: Appetite to Play +

INTERVENTIONS:
Behavioral: Appetite to Play + — In 2017 the province of BC enacted a provincial standard for physical activity, formally titled the Director of Licensing Standard of Practice - Active Play (Active Play Standards) that licensed childcare centers are required to adhere to. Along with this, a provincial capacity-building intervention (Appetite to Play) was released to provide training and education to early years providers working in the province and support the implementation of the Active Play Standards. The intervention, Appetite to Play +, will provide advanced training to early year educators on the Appetite to Play activities and resources. The intervention will include workshops and training on physical literacy, fundamental movement skills, and creating a supportive environment to sustain Active Play practices. As part of the intervention, managers will also be provided with resources to aid them with the integration of Active Play into their curriculums and schedules.

SUMMARY:
The BC government and partners developed Active Play Standards and a capacity-building strategy to help childcare centers implement the Standards. We have developed an intervention to supplement the governmental capacity-building strategies. The intervention is comprised of implementation support strategies targeted at childcare providers in BC that will aid with the sustainment of Active Play best practices at their facilities. The impact of the intervention will be assessed by measuring its impact on a) change in practices with respect to Active Play; and b) improving child-level outcomes (children's physical activity, sedentary behavior, and motor skill competencies). The findings will inform future policies and enhance our understanding of how policy action supported by communication, capacity-building, and sustainment strategies influence the environment of childcare centres.

DETAILED DESCRIPTION:
The Director of Licensing Standard of Practice - Active Play (Active Play Standard), mandates the provision of Active Play opportunities (amount of time spent outdoor, amount of physical activity, provision of fundamental skills) in licensed childcare centers in British Columbia, Canada. To support the implementation of this standard, the province released a capacity-building intervention, called Appetite to Play (ATP). Appetite to Play provides training and support to childcare providers in enhancing physical activity, physical literacy, and healthy eating environments in their facilities. To encourage the sustained use of ATP and aid childcare facilities in maintaining their adherence to the Active Play Standard, we have developed an intervention called, Appetite to Play +, targeted at facility managers and staff. The intervention builds upon ATP and is considered advanced training for childhood educators. The intervention involves the implementation of support strategies focused on integrating Active Play and fundamental movement skills into scheduling, curriculum planning, and creating a supportive environment for Active Play and healthy eating in childcare facilities.

ELIGIBILITY:
Inclusion Criteria for childcare center:

* Located in the Metro Vancouver region
* Provides care to at least 10 children older than 2 1/2 years and younger than 6 years
* Childcare program that is longer than 4 hours each day

Inclusion for child outcomes / measurement

* children must attend a childcare that has volunteered to participate in the study
* Child must be older than 2 1/2 years and younger than 6 years of age

Inclusion Criteria for managers and staff childcare centers:

- Managers at licensed BC childcare facilities, working full time (at least 3 full days per week) in a facility for children aged 2½ to 6 years, defined as an Executive Director, supervisor, or program manager. Aged 19 years or older.

OR

- Childcare staff at licensed BC childcare facilities, working full time (at least 3 full days per week), defined as Early Childhood Educator, instructor, or staff that cares for 2½ to 6-year-old children. Aged 19 years or older.

Exclusion Criteria for childcare center:

* Located outside Metro Vancouver region
* Facilities caring only for children under 2 1/2 years old or older than 6 years
* Family or in-home multi-age childcare

Exclusion Criteria for managers and staff childcare centers:

* Do not care or supervise 2 ½ to 6 years old children
* Work less than 3 full days per week
* Administrative assistant/office manager
* Younger than 19 years of age

Min Age: 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in practices related to active play (AP) and fundamental movement skills (FMS) | Two time points -baseline and 3-month post intervention
  Change in AP and FMS practices will examine child engagement in AP and FMS activities at the facility (e.g., time spent in AP, FMS, and outdoor activities, adherence to best practices). Assessment through observed practices using the Environment and Policy Assessment and Observation (EPAO) tool, and through self-reported practices based on questions developed by the Early Years Survey and the EPAO as a Self-Report instrument (EPAO-SR).
Fundamental movement skills (child outcomes) | Two time points -baseline and 3-month post intervention
  Children's FMS will be assessed with the validated Test of Gross Motor Development (TGMD-3 a norm-referenced tool for assessing 13 gross motor skills). The measure takes 15-20 min per child to administer and provides standardized and percentile composite scores for the locomotor, object control, and gross motor quotient (GMQ) composites.

SECONDARY OUTCOMES:
Characteristics of childcare settings | Three time points -baseline and 3-month, and 6-month post intervention
  Assessment of organizational processes, structural support, and processing supporting implementation of Active Play policies as measured by the Early Years Survey and the Environment and Policy Assessment and Observation as a Self-Report tool (EPAO-SR), including actions to prioritize AP and changes in the environment to support AP and FMS.
Characteristics of providers | Three time points -baseline and 3-month, and 6-month post intervention
  Assessment of staff and manager's knowledge and skills, self-efficacy, and commitment to changes facility practices to implement Active Play standards, as measured by the Early Years Survey and the EPAO-SR.

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Masse, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Masse LC, Wright C, Buckler EJ, De-Jongh Gonzalez O, Wolfenden L, Faulkner G, Carson V, Temple V, Brussoni M, Fakih S, Sauve K, Edache I, Naylor PJ. Facility-level implementation strategies in early childhood education and care to enhance adherence to a provincial physical activity standard: Protocol for the Good Start Matters ATP+ randomised controlled trial. PLoS One. 2025 Aug 12;20(8):e0329276. doi: 10.1371/journal.pone.0329276. eCollection 2025. PMID 40794716